CLINICAL TRIAL: NCT01522703
Title: Dietary Interventions and Asthma Treatment: A Pilot Study of the Effects of Whole Sprouts on Airway Allergic Inflammation
Brief Title: Effects of Whole Sprouts on Airway Allergic Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Elizabeth Matsui, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00067371; 1P01ES018176-01 (NIH)
Record Dates: First submitted 2012-01-09; First posted 2012-02-01 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-10

CONDITIONS: Allergic Rhinitis; Asthma; Allergy
Keywords: asthma; allergic rhinitis; dietary interventions; mouse allergy
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Broccoli Sprouts (Experimental): Broccoli Sprout sandwich/wrap will be eaten daily for 3 consecutive days
  Interventions: Drug: Broccoli Sprouts
- Alfalfa Sprouts (Placebo Comparator): Alfalfa Sprouts will be eaten daily in a sandwich form for 3 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Broccoli Sprouts — 100g of either broccoli or alfalfa sprouts will be eaten daily in a sandwich or wrap form.
  Other Names: sprouts, broccoli sprouts
  Arms: Broccoli Sprouts
Drug: Placebo — Alfalfa Sprouts
  Other Names: sprouts, alfalfa, broccoli sprouts
  Arms: Alfalfa Sprouts

SUMMARY:
The primary objective of this study is to determine if broccoli sprouts (BS) improves airway inflammatory, oxidative stress (OS), and symptoms among asthmatic adults with aeroallergen sensitization.

The study is a double-blind, placebo-controlled, randomized trial to compare BS to placebo in 40 adults with asthma. 40 adults (age 18-50) who meet these eligibility criteria will be randomized to receive either: (a) BS or (b) placebo (alfalfa sprouts). Subjects will eat a sprouts sandwich daily for three days, and then undergo repeat measurement of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* doctor diagnosis of asthma
* aeroallergen sensitization
* Non-smoker
* Negative pregnancy test
* Not breastfeeding
* Normal TSH
* For women, abstinent or using reliable birth control
* Age 18-50 years
* No other major pulmonary disease such as cystic fibrosis or COPD
* Willingness to participate in study and sign consent form

Exclusion Criteria:

* Severe or unstable asthma defined as requiring hospitalization in the previous 6 months or intubation in the previous 2 years, or on high-dose inhaled corticosteroids or chronic oral corticosteroids
* Uncontrolled asthma defined as short-acting beta agonist use 3 or more days a week in the previous 4 weeks
* Other significant medical issues such as heart disease or poorly controlled hypertension, type 1 diabetes, poorly controlled type 2 diabetes, or hypothyroidism
* Pregnancy or nursing/breastfeeding mothers
* On beta-blocker therapy
* On reserpine, clonidine, imipramine, or related tricyclic drugs
* Taking anti-oxidant supplements
* Planned dietary changes during the study period
* Unable to stop antihistamines prior to skin testing
* Food allergy to Broccoli Sprouts or Alfalfa Sprouts
* Omalizumab use within the last 12 months
* Nasal polyps

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Matsui, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Broccoli Sprouts: ingestion of broccoli sprouts 3 consecutive days
- Alfalfa Sprouts (Placebo Control): ingestion of alfalfa sprouts 3 consecutive days
Period: Overall Study
Arm/Group | Broccoli Sprouts | Alfalfa Sprouts (Placebo Control)
Started | 25 | 26
Completed | 20 | 20
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Broccoli Sprouts | Alfalfa Sprouts (Placebo Control) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (9.6) | 34.2 (9.2) | 33.6 (9.4)
Gender [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Nitric Oxide Concentrations
Description: exhaled nitric oxide concentrations
Time Frame: at 3 days
Measure: Median (Inter-Quartile Range); unit: ppb
Groups:
- Alfalfa Sprouts (Placebo Control): ingestion of alfalfa sprouts for 3 consecutive days
- Broccoli Sprouts: ingestion of broccoli sprouts for 3 consecutive days
Arm/Group | Alfalfa Sprouts (Placebo Control) | Broccoli Sprouts
Number analyzed (Participants) | 20 | 20
ppb | 22 [12 to 32] | 19 [15 to 43]

ADVERSE EVENTS:
Arm/Group | Broccoli Sprouts | Alfalfa Sprouts (Placebo Control)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No